CLINICAL TRIAL: NCT01996319
Title: MOVE - A Randomized, Double-blind, Placebo-controlled, Multicenter, Cross-over Study to Assess the Effects of a 3 Week Therapy Each With QVA149 Versus Placebo on Pulmonary Function and Average Physical Activity Levels in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Randomized, Double-blind, Placebo-controlled, Multicenter, Cross-over Study to Assess the Effects of a 3 Week Therapy Each With QVA149 Versus Placebo on Pulmonary Function and Average Physical Activity Levels in Patients With COPD.
Acronym: MOVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149ADE03
Record Dates: First submitted 2013-11-15; First posted 2013-11-27 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Treatment sequence I (Active Comparator): QVA149 once a day during 21 days cross-over to placebo once a day for up to 21 days
  Interventions: Drug: QVA149; Drug: Placebo
- Treatment sequence II (Active Comparator): Placebo once a day during 21 days cross-over to QVA149 once a day for 21 days
  Interventions: Drug: QVA149; Drug: Placebo

INTERVENTIONS:
Drug: QVA149 — QVA149 (110/50 µg) once a day via Breezhaler® device
Drug: Placebo — Placebo once a day via Breezhaler® device

SUMMARY:
This study is designed to assess the effect of QVA149 (110/50 ug q.d.) versus placebo on pulmonary function and average physical activity levels in patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

Patients with stable COPD according to the current GOLD guidelines (GOLD 2013). Current or ex-smokers who have a smoking history of at least 10 pack years (e.g. 10 pack years = 1 pack /day x 10 yrs, or ½ pack/day x 20 yrs)..

Patients with airflow limitation indicated by a post-bronchodilator FEV1 ≥40% and <80% of the predicted normal, and a post-bronchodilator FEV1/FVC <0.70

Exclusion Criteria:

Patients with conditions contraindicated for treatment with, or having a history of reactions/hypersensitivity to any of the following inhaled drugs, drugs of a similar class or any component thereof, anticholinergics, long and short acting beta2 agonists, sympathomimetic amines, lactose or any of the other excipients Patients who have a clinically significant ECG abnormality at Visit 1, who in the judgment of the investigator would be at potential risk if enrolled into the study.

Patients with paroxysmal (e.g. intermittent) atrial fibrillation are excluded. Patients with persistent atrial fibrillation as defined by continuous atrial fibrillation for at least 6 months and controlled with a rate control strategy (i.e., beta blocker, calcium channel blocker, pacemaker placement, digoxin or ablation therapy) for at least 6 months may be considered for inclusion. In such patients, atrial fibrillation must be present at baseline and screening visits, with a resting ventricular rate < 100/min.

Patients with Type I or uncontrolled Type II diabetes and patients with a history of blood glucose levels consistently outside the normal range Patients with narrow-angle glaucoma, symptomatic prostatic hyperplasia or bladder-neck obstruction or moderate to severe renal impairment or urinary retention.

Patients with a history of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin. Patients with non-melanoma skin carcinoma may be considered for the study.

Patients with a body mass index (BMI) of more than 40 kg/m2. Women who are pregnant or breast feeding Patients requiring long term oxygen therapy on a daily basis for chronic hypoxemia.

Patients who have had a COPD exacerbation that required treatment with antibiotics and/or oral corticosteroids and/or hospitalization in the 6 weeks prior to screening.

Patients who have had a respiratory tract infection within 4 weeks prior to screening.

Patients with any history of asthma. Patients with concomitant pulmonary disease Patients with clinically significant bronchiectasis. Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- Germany (27):
  - Novartis Investigative Site, Heidelberg, Germany
  - Novartis Investigative Site, Potsdam, Germany
  - Novartis Investigative Site, Teterow, Germany
  - Novartis Investigative Site, Koblenz, North Rhine-Westphalia
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Geesthacht, Schleswig-Holstein
  - Novartis Investigative Site, Berlin, State of Berlin
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düren
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Euskirchen
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Höchstadt an der Aisch
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rheine
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Wiesloch

REFERENCES:
- [Derived] Watz H, Mailander C, Baier M, Kirsten A. Effects of indacaterol/glycopyrronium (QVA149) on lung hyperinflation and physical activity in patients with moderate to severe COPD: a randomised, placebo-controlled, crossover study (The MOVE Study). BMC Pulm Med. 2016 Jun 14;16(1):95. doi: 10.1186/s12890-016-0256-7. PMID 27301417

RESULTS

PARTICIPANT FLOW:
Groups:
- QVA149 Then Placebo: QVA149 once a day during 22 days cross-over to placebo once a day for up to 22 days
- Placebo Then QVA149: Placebo once a day during 22 days cross-over to QVA149 once a day for 22 days
Period: Overall Study
Arm/Group | QVA149 Then Placebo | Placebo Then QVA149
Started | 96 | 98
Completed | 88 | 95
Not Completed | 8 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Severe or moderate (COPD) Exacerbation | 5 | 1
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 Then Placebo | Placebo Then QVA149 | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (7.9) | 61.2 (7.7) | 62.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 67
  Male | 64 | 63 | 127

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Inspiratory Capacity (IC) Comparison Between QVA149 and Placebo
Description: Inspiratory capacity (IC) will be measured with spirometry conducted according to internationally accepted standards. The mean of 3 acceptable measurements will be calculated and reported in liters. In this cross-over trial, we had two baselines collected at day 1 and collected at day 36. From the IC measurements collected on either Day 22 or 57, respectively, the appropriate baseline measurements were subtracted - so either Day 22-Day1 or Day 57-Day36
Time Frame: Baseline, day 22, baseline day 36, day 57
Population: Full Analysis Set (FAS): all randomized patients who applied at least one dose of study medication during at least one study period. all patients were included in these analyses when baseline and day 22 data plus baseline day 36 and day 57 data were available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 189 | 184
Liters | 0.3790 (0.2747) [0.3464 to 0.4117] | 0.1769 (0.1933) [0.1379 to 0.2159]
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; null hypoth = 0.2021, 95% CI 2-sided [0.1583 to 0.2460]

2. Primary Outcome: Change From Baseline in the Comparison of QVA149 Versus Placebo With Respect to Average Physical Activity Level
Description: Average physical activity level is defined by average daily activity-related energy consumption [Kcal/day], measured via Actinography device. In this cross-over trial, we had two baselines collected at day 1 and collected at day 36. From the activity measurements collected on either Day 22 or 57, respectively, the appropriate baseline measurements were subtracted - so either Day 22-Day1 or Day 57-Day36
Time Frame: Baseline, day 22, baseline day 36, day 57
Population: Full Analysis Set (FAS): all randomized patients who applied at least one dose of study medication during at least one study period. Only patients with baseline and day 22 data, plus baseline on day 36 and day 57 data were included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: kcal/day
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 175 | 170
kcal/day | 5.1063 (214.6) [-24.4000 to 34.6125] | -31.6063 (233.0) [-61.5268 to -1.6857]
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority or Other; p = 0.0399, ANCOVA; Null hypoth = 36.7126, 95% CI 2-sided [1.7241 to 71.7011]

3. Secondary Outcome: Change in the Comparison of QVA149 vs. Placebo on the Average Number of Steps Per Day
Description: The average number of steps per day will be measured via Actinography device. In this cross-over trial, we had two baselines collected at day 1 and collected at day 36. From the activity measurements collected on either Day 22 or 57, respectively, the appropriate baseline measurements were subtracted - so either Day 22-Day 1 or Day 57-Day36
Time Frame: Baseline, day 22, baseline day 36, day 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Steps/day
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 178 | 173
Steps/day | 30.7 (1662) | -320.7 (1648)

4. Secondary Outcome: Change in the Duration of at Least Moderate Activity Per Day Comparison of QVA149 Versus Placebo
Description: Least moderate activity (defined as 3,5-7kcal/min) will be measured via Actinography device. In this cross-over trial, we had two baselines collected at day 1 and collected at day 36. From the activity measurements collected on either Day 22 or 57, respectively, the appropriate baseline measurements were subtracted - so either Day 22-Day1 or Day 57-Day36
Time Frame: Baseline, day 22, baseline day 36, day 57
Population: Full Analysis Set (FAS): all randomized patients who applied at least one dose of study medication during at least one study period. Only patients with baseline and day 22, plus baseline day 36 and day 57 data were included in this analysis.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 178 | 173
Minutes | -5.5 (51.8) | -13.0 (52.3)

5. Secondary Outcome: Change From Baseline in Peak IC Comparison Between QVA149 and Placebo on Day 1.
Description: Inspiratory capacity (IC) will be measured with spirometry conducted according to internationally accepted standards. The mean of 3 acceptable measurements will be calculated and reported in liters. In this cross-over trial, we had two baselines collected at day 1 and collected at day 36. The IC measurements collected prior to dosing on either Day 1 or 36, respectively, were subtracted from the appropriate peak measures on the same respective days
Time Frame: Day 1 or day 36
Population: Full Analysis Set (FAS): all randomized patients who applied at least one dose of study medication during at least one study period. Only patients with baseline and day 1 post treatment initiation were included in this analysis.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 193 | 186
Liters | 0.486 (0.2752) | 0.207 (0.2114)

6. Secondary Outcome: Change From Baseline in the Trough IC Comparison Between QVA149 and Placebo
Description: as for outcome 1
Time Frame: Baseline, day 22, baseline day 36, day 57
Population: Full Analysis Set (FAS): all randomized patients who applied at least one dose of study medication during at least one study period. Only patients with baseline and day 20 post treatment initiation were included in this analysis.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 190 | 183
Liters | 0.210 (0.346) | -0.035 (0.279)

7. Secondary Outcome: Peak Forced Expiratory Volume 1 (FEV1) Comparison Between QVA149 and Placebo at Day 1
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The mean of 3 acceptable measurements will be calculated and reported in liters. In this cross-over trial, we had two baselines collected at day 1 and collected at day 36. The FEV1 measurements collected prior to dosing on either Day 1 or 36, respectively, were subtracted from the appropriate peak measures on the same respective days
Time Frame: Day 1 or day 36
Population: Full Analysis Set (FAS): all randomized patients who applied at least one dose of study medication during at least one study period
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 192 | 186
Liters | 0.347 (0.176) | 0.111 (0.179)

8. Secondary Outcome: Trough FEV1 Comparison Between QVA149 and Placebo After 22 Days
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The mean of 3 acceptable measurements will be calculated and reported in liters. In this cross-over trial, we had two baselines collected at day 1 and collected at day 36. From the FEV1 measurements collected on either Day 22 or 57, respectively, the appropriate baseline measurements were subtracted - so either Day 22-Day1 or Day 57-Day36
Time Frame: Baseline, day 22, baseline day 36, day 57
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 188 | 183
Liters | 0.245 (0.221) | -0.058 (0.207)

ADVERSE EVENTS:
Arm/Group | QVA149 Then Placebo | Placebo Then QVA149
Serious Adverse Events (participants affected / at risk) | 4/193 | 2/188
Other Adverse Events (participants affected / at risk) | 27/193 | 19/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 Then Placebo (N=193) | Placebo Then QVA149 (N=188)
Myocardial infarction (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 Then Placebo (N=193) | Placebo Then QVA149 (N=188)
Fatigue (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 7 | 8
Rhinitis (Infections and infestations) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Headache (Nervous system disorders) | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety